CLINICAL TRIAL: NCT00155896
Title: Establishing the Incidences of BRCA1 and BRCA2 Mutation by Combining DHPLC and Direct Sequencing in Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261700719
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2002-09

CONDITIONS: Ovarian Cancer
Keywords: BRCA1 gene, BRCA2 gene, DHPLC, genetic diagnosis
MeSH Terms: conditions — Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Ovarian cancer is the first mortality rate of gynecologic malignancies. The incidence of ovarian cancer increased in recent 10 years. Ovarian cancer indeed is a disease that should be respected, however, there were only few of research work focusing on it in Taiwan.

To study the mechanisms of carcinogenesis of ovarian cancer will help us understand this disease and develop new strategies of diagnosis and prevention for ovarian cancer in the future. The present diagnostic methods of malignancy are clinical symptoms, physical examination, evaluation of tumor markers and instruments. It is a important issue to diagnose cancer earlier to improve the survival of cancer patients. By the development of biomedical science, many genes have been identified to be related with the carcinogenesis. If we can detect the possibility of genetic mutation earlier, we may deal with the suspected areas of malignancy as soon as possible. To our present knowledge, carcinogenesis of ovarian cancer has strong correlation with some special genes such as BRCA1 and BRCA2 genes. There is 1 out of 200 normal population with BRCA1 or BRCA2 gene mutation in the western countries. The incidences of BRCA1 or BRCA2 gene mutation even increase to 30-50% in the population of familial ovarian cancer. Women with BRCA1 gene mutation have 80% to get breast cancer before the age of 70 and 63% of them would get ovarian cancer before the age of 70. Women with BRCA2 gene mutation have 80% to get breast or ovarian cancer before the age of 70. It seems that the genetic diagnosis of BRCA1/BRCA2 has its clinical practice. The development of new instrument- denaturing high-performance liquid chromatography (DHPLC) is to use automated detection to find out the minute or single mutation of nucleotide. It has been applied to the clinical service by utilizing DHPLC for the genetic diagnosis of BRCA1 and BRCA2 of breast cancer patients in the department of Genetic Medicine of our hospital. It will become a most powerful tool to establish the database of BRCA1 or BRCA2 gene mutation of the ovarian cancer patients in Taiwan, when we can use the technique of DHPLC combining with the direct DNA sequencing.

DETAILED DESCRIPTION:
Malignancy is the first cause of death in Taiwan. There are around 30,000 people died due to malignancy every year. Ovarian cancer is the first mortality rate of gynecologic malignancies. The incidence of ovarian cancer increased in recent 10 years. Ovarian cancer indeed is a disease that should be respected, however, there were only few of research work focusing on it in Taiwan.

To study the mechanisms of carcinogenesis of ovarian cancer will help us understand this disease and develop new strategies of diagnosis and prevention for ovarian cancer in the future. The present diagnostic methods of malignancy are clinical symptoms, physical examination, evaluation of tumor markers and instruments. It is a important issue to diagnose cancer earlier to improve the survival of cancer patients. By the development of biomedical science, many genes have been identified to be related with the carcinogenesis. If we can detect the possibility of genetic mutation earlier, we may deal with the suspected areas of malignancy as soon as possible. To our present knowledge, carcinogenesis of ovarian cancer has strong correlation with some special genes such as BRCA1 and BRCA2 genes. There is 1 out of 200 normal population with BRCA1 or BRCA2 gene mutation in the western countries. The incidences of BRCA1 or BRCA2 gene mutation even increase to 30-50% in the population of familial ovarian cancer. Women with BRCA1 gene mutation have 80% to get breast cancer before the age of 70 and 63% of them would get ovarian cancer before the age of 70. Women with BRCA2 gene mutation have 80% to get breast or ovarian cancer before the age of 70. It seems that the genetic diagnosis of BRCA1/BRCA2 has its clinical practice. The development of new instrument- denaturing high-performance liquid chromatography (DHPLC) is to use automated detection to find out the minute or single mutation of nucleotide. It has been applied to the clinical service by utilizing DHPLC for the genetic diagnosis of BRCA1 and BRCA2 of breast cancer patients in the department of Genetic Medicine of our hospital. It will become a most powerful tool to establish the database of BRCA1 or BRCA2 gene mutation of the ovarian cancer patients in Taiwan, when we can use the technique of DHPLC combining with the direct DNA sequencing.

So we propose this research project. There are two main purposes in this project. First, we will utilize the new technique of DHPCL with direct DNA sequence to set up the database of BRCA1 and BRCA2 gene mutation of ovarian cancer patients in Taiwan. We can screen out BRCA1 and BRCA2 gene mutation from high-risk group by this new technique. And then we can provide these patients suitable genetic consulting and related treatment planning. Second, we would lie to set up the new technique of DHPLC combining with direct DNA sequencing in the genetic diagnosis of ovarian cancer patients for the future clinical service in our hospital.

ELIGIBILITY:
Inclusion Criteria:

- ovarian cancer

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-01; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan